CLINICAL TRIAL: NCT05921890
Title: To Evaluate the Safety and Tolerability of GS3-007a Oral Solution in a Multi-dose, Randomized, Open, Single-center Study in Healthy Chinese Adult Subjects.
Brief Title: To Evaluate the Safety and Tolerability of Multiple Doses of GS3-007a Oral Solution in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GenSci073-104
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-06

CONDITIONS: Healthy Subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GS3-007 oral liquid (Experimental): 36 subjects，12 subjects in each dose group. Two dose groups were planned: 0.8 mg/kg and 1.6 mg/kg once a day for 4 weeks. According to the research progress of 1.6mg/kg QD, it was decided whether to add 0.8 mg/kg twice a day for 4 weeks.
  Interventions: Drug: GS3-007 oral liquid

INTERVENTIONS:
Drug: GS3-007 oral liquid — The dosage was calculated according to body weight, once a day or twice a day.

SUMMARY:
To evaluate the safety and tolerability of GS3-007a oral solution after multiple oral administration in Chinese healthy adult subjects.

DETAILED DESCRIPTION:
To evaluate the pharmacodynamic (PD) and pharmacokinetics（PK） characteristics of GS3-007a oral solution after multiple oral administration in Chinese healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects aged 18-45 years (including boundary values), male or female;
* Body mass index: 19-26 kg/m2 (including boundary values), male weight ≥50 kg, female weight ≥45 kg;

Exclusion Criteria:

* (Screening period consultation) accumulated two or more allergies to other drugs, food and environment; Or prone to rash, urticaria and other allergic symptoms; Or are known to be allergic to growth hormone-promoting peptide drugs or excipients of this preparation;
* (screening period) have a clear history of neurological or mental disorders; Persons with incapacity or cognitive impairment;
* ALT and AST exceed the upper limit of the normal range;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
TEAEs | 35 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital Affiliated to North Sichuan Medical College, Chengdu, Sichuan, China